CLINICAL TRIAL: NCT02149823
Title: Examining Dose-Related Effects of Oxytocin on Social Cognition Across Populations
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: All study proceedings stopped prematurely due to Covid-19 restrictions for intranasal formulations
Sponsor: Maria de las Mercedes Perez Rodriguez (Other)
Collaborators: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency); VISN 3 Mental Illness Research, Education and Clinical Center (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Maria de las Mercedes Perez Rodriguez, Fellow, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: GCO 13-0340; UL1TR000067 (NIH)
Record Dates: First submitted 2014-05-21; First posted 2014-05-29 (Estimated); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Borderline Personality Disorder; BPD; Schizotypal Personality Disorder; SPD; Autism Spectrum Disorder; Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
Keywords: Oxytocin, Social Cognition; Borderline Personality Disorder; Schizotypal Personality Disorder; Social Cognition; BPD; SPD; MASC; Autism Spectrum Disorder; Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
MeSH Terms: conditions — Borderline Personality Disorder; Schizotypal Personality Disorder; Autism Spectrum Disorder; Schizophrenia; Psychotic Disorders; Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Intranasal Oxytocin Group 1 (Active Comparator): Placebo on visit 1, oxytocin 24IU on visit 2, then 40 IU on visit 3
  Interventions: Drug: Syntocinon 24 Intranasal Units (IU); Drug: Syntocinon 40 Intranasal Units (IU); Drug: Intranasal Placebo
- Intranasal Oxytocin Group 2 (Active Comparator): oxytocin 24IU on visit 1, placebo on visit 2, then oxytocin 40IU on visit 3
  Interventions: Drug: Syntocinon 24 Intranasal Units (IU); Drug: Syntocinon 40 Intranasal Units (IU); Drug: Intranasal Placebo
- Intranasal Oxytocin Group 3 (Active Comparator): oxytocin 40IU on visit 1, oxytocin 24IU on visit 2, then placebo on visit 3.
  Interventions: Drug: Syntocinon 24 Intranasal Units (IU); Drug: Syntocinon 40 Intranasal Units (IU); Drug: Intranasal Placebo
- Intranasal Oxytocin Group 4 (Active Comparator): after visit 4, placebo on subsequent visit , then oxytocin 40IU at following visit
  Interventions: Drug: Syntocinon 40 Intranasal Units (IU); Drug: Intranasal Placebo
- Intranasal Oxytocin Group 5 (Active Comparator): after visit 4, oxytocin 40IU on subsequent visit, then placebo at following visit
  Interventions: Drug: Syntocinon 40 Intranasal Units (IU); Drug: Intranasal Placebo

INTERVENTIONS:
Drug: Syntocinon 24 Intranasal Units (IU)
  Other Names: Intranasal Oxytocin
  Arms: Intranasal Oxytocin Group 1; Intranasal Oxytocin Group 2; Intranasal Oxytocin Group 3
Drug: Syntocinon 40 Intranasal Units (IU)
  Other Names: Intranasal Oxytocin
Drug: Intranasal Placebo

SUMMARY:
Social cognition impairment is critical to the pathology and morbidity of a number of psychiatric disorders, including the schizophrenia spectrum, the autism spectrum and the personality disorders, thus representing a dimension consistent with RDoC. As such, this study aims to a) further characterize the unique deficits in social cognition (recognition and interpretation of social cues and representation of thoughts, intentions, and feelings of others) across disorders, including the schizophrenia spectrum (which includes schizophrenia, SCZ, schizoaffective disorder, SAD, bipolar disorder, BD, and schizotypal personality disorder, SPD), the autism spectrum disorders (ASD), and borderline personality disorder (BPD) compared to healthy controls (HC); b) assess the effect of intranasal oxytocin (OXT) as a regulator and novel treatment of social cognition impairment in these disorders; and c) enhance our understanding of the specificity and exact mechanisms of impairment to inform the accurate dosing of OXT required to modulate social cognition in these disorders and identify a model of optimum social cognitive function. Addressing these questions will further catalyze research into a model of optimum social cognitive activity, and accelerate industry development of agents suited to routine clinical administration.

DETAILED DESCRIPTION:
Social cognitive impairments, particularly deficits and distortions in recognition and interpretation of social cues and representations of thoughts, intentions, and feelings of others-termed mentalization-are a key contributor to the pathology and morbidity of a number of psychiatric disorders, including the schizophrenia spectrum, the autism spectrum and personality disorders. Individuals with schizophrenia spectrum disorders have deficits in social cognition (hypomentalization), while individuals with borderline personality disorder seem to have exaggerated and distorted social cognition (hypermentalization). However, the specificity and mechanisms of these impairments remain unclear. Therefore, a better understanding of the modulation of social cognition is a priority for developing interventions both pharmacologic and psychosocial. We propose here to examine the effects of oxytocin, known to be a key regulator of social cognition through modulating frontolimbic neural circuitry, on social cognition in schizotypal and borderline patients. In doing so, we aim to characterize a model of optimum social cognitive activity to direct the development of treatments, including dosing and target population-specific effects.

To this end, we propose to perform a 2-year study in which 105 patients, (45 with schizophrenia spectrum disorders, 30 with borderline personality disorder, and 30 with autism spectrum disorders) will perform 3 rounds of social cognition testing after three acute single-dose treatment conditions (intranasal oxytocin dose of 24IU or 40IU or placebo) separated by a washout period, in a repeated-measures, within-subjects, randomized, placebo-controlled, double-blind, counterbalanced cross-over proof-of concept design. 30 healthy controls will not receive oxytocin/placebo and will perform 3 rounds of social cognition tests separated by approximately 4 weeks, serving as a benchmark for normal performance and a control for practice effects. Social cognitive testing will be performed 45 minutes after drug/placebo administration in an identical protocol each time. The social cognitive test serving as primary outcome measure will be the Movie for the Assessment of Social Cognition (MASC). We will also include other tests of social cognition and symptom measures, to evaluate scope of effects. We will compare outcome measures at baseline (placebo day) in schizotypal and borderline patients and healthy controls, and in schizotypal and borderline patients across drug doses and placebo administration.

Furthermore, 60 subjects (15 HC, 15 with schizophrenia spectrum disorders, 15 BPD, and 15 with autism spectrum disorders, either new subjects or already enrolled subjects) will be expected to complete an add-on MRI component of the study, after signing an additional consent form. For the MRI portion of the study, these subjects will perform 2 more rounds of social cognition testing after receiving double-blind intranasal oxytocin (40 IU) or placebo in randomized order, in a cross-over, within-subjects design, separated by approximately a 1-week washout. The subjects will receive the study medication directly prior to beginning an fMRI scan that will last approximately two hours. Oxytocin levels will be measured before oxytocin administration and every 10-15 minutes until about 2 hours and 30 minutes post-administration. The remainder of the protocol will remain the same.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ age ≤ 65
* Medically and neurologically healthy
* Willing and able to provide informed consent
* IQ≥80

Exclusion Criteria:

* Currently meets for a psychotic episode
* Clinically significant cardiovascular or neurological conditions, traumatic brain injury, uncontrolled hypertension, clinically significant EKG abnormalities, or serious general medical illness
* Clinical evidence of dehydration or significant hypotension; pregnant or lactating
* Currently meets DSM-IV-TR criteria for MDD
* Current substance abuse (last 6 months) or past dependence on stimulants, opioids or other potentially neurotoxic drugs
* Currently taking psychotropic or other systemic medications
* Non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-09; Primary Completion 2020-07 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Movie for the Assessment of Social Cognition (MASC) | Day 1
  The MASC involves watching a 15 min movie about 4 characters getting together for a dinner party. The video is paused 45 times and questions concerning the characters' feelings, thoughts, and intentions are asked. It takes 40 min to complete. The multiple choice version of the MASC allows a qualitative social cognition error analysis.
Movie for the Assessment of Social Cognition (MASC) | Day 29
Movie for the Assessment of Social Cognition (MASC) | Day 57

SECONDARY OUTCOMES:
Reading of the Mind in the Eyes | Day 1
  The 'Reading the Mind in the Eyes' (Eyes) test is an advanced test of theory of mind. It is widely used to assess individual differences in social cognition and emotion recognition across different groups and cultures. The social cognition measure will be administered as a control task.
Reading of the Mind in the Eyes | Day 29
Reading of the Mind in the Eyes | Day 57
Resting-state functional connectivity | Day 1
  Participants will undergo resting-state functional MRI scanning while viewing a fixation cross on a black screen, with instructions to lie still and keep their eyes open. A non-invasive eye-tracking device (available as an MRI peripheral) will be used to ensure that participants do not fall asleep during the long resting-state period, and to track eye gaze during the social cognition task. Resting-state scanning will be done during the onset of oxytocin effects until peak effects are achieved (approximately 30 minutes post administration)
Resting-state functional connectivity | Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Maria de las Mercedes Perez Rodriguez, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; James J. Peters VA Medical Center
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - James J Peters VA Medical Center, The Bronx, New York